CLINICAL TRIAL: NCT01444105
Title: A Prospective, Randomized, Controlled, Parallel Groups Evaluation of Open-angle Glaucoma Subjects on One Ocular Hypotensive Medication Randomized to Treatment With Two Trabecular Micro-bypass Stents or Selective Laser Trabeculoplasty
Brief Title: Open-angle Glaucoma Subjects on One Ocular Hypotensive Medication Randomized to Treatment With Two Trabecular Micro-bypass Stents or Selective Laser Trabeculoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCF-028
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Open-angle Glaucoma
Keywords: Open angle glaucoma; Pseudoexfoliative glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- iStent (Active Comparator): implantation of two iStent devices
  Interventions: Device: iStent
- SLT (Active Comparator): Laser treatment
  Interventions: Other: SLT

INTERVENTIONS:
Device: iStent — Implantation of two iStent devices
  Arms: iStent
Other: SLT — Laser treatment
  Arms: SLT

SUMMARY:
Evaluation of intraocular pressure (IOP) lowering effect of two iStent stents versus a SLT procedure in subjects with open-angle glaucoma on one ocular hypotensive medication.

DETAILED DESCRIPTION:
Evaluation of intraocular pressure (IOP) lowering effect of two iStent stents versus a SLT procedure in subjects with open-angle glaucoma on one ocular hypotensive medication.

ELIGIBILITY:
Inclusion Criteria:

* Phakic study eye or study eye with a posterior chamber intraocular lens (PC-IOL)
* Primary open-angle glaucoma (including pseudoexfoliative)

Exclusion Criteria:

* Aphakic or pseudophakic with anterior chamber IOLs (AC-IOLs) (study eye)
* Prior stent implantations (study eye)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean diurnal IOP (mm Hg) at the Month 12 visit. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Lilit A Voskanyan, MD, PhD, Principal Investigator — S.V. Malayan Ophthalmological Center, Yerevan, Armenia
Locations (1):
- S.V. Malayan Ophthalmological Center, Yerevan, Armenia

REFERENCES:
- [Derived] Rolim-de-Moura CR, Paranhos A Jr, Loutfi M, Burton D, Wormald R, Evans JR. Laser trabeculoplasty for open-angle glaucoma and ocular hypertension. Cochrane Database Syst Rev. 2022 Aug 9;8(8):CD003919. doi: 10.1002/14651858.CD003919.pub3. PMID 35943114